CLINICAL TRIAL: NCT04816825
Title: Feasibility and Effectiveness of a Home Monitored Rehabilitation Intervention Using an Exergaming Approach in COPD Patients - a Randomized, Controlled Clinical Study
Brief Title: Home-monitored Telerehabilitation in COPD Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ExerGaming
Record Dates: First submitted 2021-03-18; First posted 2021-03-25 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-03

CONDITIONS: Copd
Keywords: COPD; Telerehabilitation; Pulmonary rehabilitation; exergaming
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: A randomized clinical controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exergaming (Experimental): The combination of 1) game-console based exercise programs, 2) specifically designed by professional physiotherapists with focus on subjects with a chronic lung disease and 3) weekly distant monitoring with close supervision by a physiotherapist. Individually prescribed exercise program based on tests of patient's physical fitness.
  Interventions: Device: Alkit eSence
- Standard rehabilitation (Active Comparator): Standard rehabilitation at the COPD-Center. This includes recommendations about physical activity according to the general guidelines, however, individualized after each subject's physical fitness level.
  Interventions: Other: Standard rehabilitation

INTERVENTIONS:
Device: Alkit eSence — Home-based rehabilitation program including computer games and supervised by a physiotherapist.
  Arms: Exergaming
Other: Standard rehabilitation — Standard rehabilitation program at the COPD-Center
  Arms: Standard rehabilitation

SUMMARY:
Study title Feasibility and effectiveness of a home monitored rehabilitation intervention using an exergaming approach in COPD patients - a randomized, controlled study.

Background and rationale Chronic Obstructive Pulmonary Disease (COPD) is a common chronic disease characterized by persistent airflow limitation caused by significant exposure to noxious particles or gases, particularly cigarette smoking. In Sweden the prevalence of COPD is approximately 8% and the annual estimated cost for society of 9.1 billion SEK. Improving exercise capacity and physical activity levels are important goals in management of patients with COPD and are strong determinants of positive outcomes, including increased quality of life. Major barrier for rehabilitation recommendations is the limited access and adherence to organized center-based exercise programs. Major barriers related to the side of health care organization are budgets and infrastructure and the limitation in time of the programs. From patient's perspective major barriers exist, like distance, and lack of transport to the unit, also in relation to the frequency of the program, which is commonly two times a week.

Research question and objectives The primary objective of this study is to investigate whether home-based telemonitored supervised exercise programs using an exergaming approach will be associated to improved physical fitness, measured with the (1-minute sit-to-stand test, 1-MSTST) compared to the ordinary care.

The secondary objectives of this study are:

1. To investigate whether a home-based exergaming program is associated with improved health-related quality of life, exercise capacity, physical activity levels and body composition.
2. To investigate if the home-based exergaming program is associated with less exacerbations.
3. To investigate if the home-based exergaming program is associated with improved health care utilization and/or less hospitalization from all causes?

Study design This is an open label , randomized controlled clinical study. The study takes place at the COPD-center at Sahlgrenska University hospital. Subjects will be randomized to either the use of the ALKIT exergaming tool in combination with telemonitored supervision by a physiotherapist or ordinary care without this system at their first visit. A total of 92 subjects will be included in the study, 46 in every arm. The intervention will include exergames performed 3 times a week for 12 weeks, consistent with the current recommendations. Pre-and post-intervention tests will be performed and subjects in both groups will be assessed. The tests include: 1-minute sit-to-stand test, 6-minute walk test, and timed-up and go. Two self- assessed questionnaires will be filled in: COPD Assessment Test and EQ5D-5L. Subjects will be also measured for quadriceps muscle strength, shoulder flexion and body composition. Additionally, physical activity level will be assessed by outcomes of pedometer worn over a week. Moreover, exacerbations and health care utilization will be measured. Users' perception of the exergaming program will be also investigated.

Population and study size The study will include a total of 92 subjects, 46 in the intervention- and 46 in the control arm. For each participant, the total study participation time will be 12 weeks. A randomization list will be produced with random assignment of treatment groups in a ratio of 1:1

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to participate and signed informed consent form
2. Diagnosis of COPD
3. FEV1/FVC (post bronchodilator) <0.7
4. GOLD severity grade B/D
5. FEV, < 80% predicted
6. Cognitive ability relevant for the studies as judged by the investigator
7. Living in their own home and able to manage their activities of daily living

Exclusion Criteria:

1. Rapidly progressing severe disease other than COPD and COPD-related diseases.
2. Influencing the HRQOL during the study time as judged by the investigator, e.g. long-term stay (>2 weeks) away from home during the study period.
3. Inability to communicate in Swedish.
4. Any condition that may interfere with the possibility for the subject to comply with the study protocol.
5. Already participating in the pulmonary rehabilitation training group 2 times a week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Physical activity | Baseline and 12 weeks after baseline
  Change in level of physical activity will be objectively measured with 1-minute sit to stand test

SECONDARY OUTCOMES:
Exercise capacity | Baseline and 12 weeks after baseline
  Change in submaximal exercise capacity will be measured by 6-Minute Walking Test.
Exercise capacity | Baseline and 12 weeks after baseline
  Change in submaximal exercise capacity will be measured by Timed up and go (TUG) test.
Exercise capacity | Baseline and 12 weeks after baseline
  Change in submaximal exercise capacity will be assessed by outcomes of a pedometer (number of daily steps).
Body composition | Baseline and 12 weeks after baseline
  Change in body composition will be calculated by Body Mass Index (BMI) by a BIA device.
Body composition | Baseline and 12 weeks after baseline
  Change in body composition will be calculated by Fat Free Mass Index (FFMI) by a BIA device.
Body strength | Baseline and 12 weeks after baseline
  Change in quadriceps muscle strength measured by the One-Repetition Maximum test (1RM). Muscle endurance will be measured by a shoulder flexion test (SFT).
Body strength | Baseline and 12 weeks after baseline
  Change in muscle endurance will be measured by a shoulder flexion test (SFT).
Health-related quality of life | Baseline and 12 weeks after baseline
  Change in disease-specific quality of life by using a COPD Assessment Test (CAT) questionnaire. CAT measures COPD symptoms with scores from 0 to 5 points (0 indicating no impact or symptoms, 5- worst possible impact or symptoms) summing up to a total CAT score range of 0-40 points.
Health-related quality of life | Baseline and 12 weeks after baseline
  Change in general health-related quality of life will be measured by The 5-level EQ-5D EuroQoL (EQ5D-5L) questionnaire. First part of the questionnaire indicates health state in 5 dimentions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The total score ranges 5-25 and higher score indicates worse health condition. The second part of EQ5D-5L, the EQ VAS (Visual Analog Score) records the patient's self-rated health on a vertical visual analogue scale (0-100), where the endpoints are labelled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0). This part will be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Number of exacerbations | Baseline and 12 weeks after baseline
  Change in exacerbation incidence will be measured by number of courses of corticosteroids and/or antibiotics for a worsening of respiratory symptoms.
Healthcare utilization | Baseline and 12 weeks after baseline
  Change in healthcare utilization will be measured by number of hospital admissions for COPD.
Healthcare utilization | Baseline and 12 weeks after baseline
  Change in healthcare utilization will be measured by number of hospital admissions for all causes.

OTHER OUTCOMES:
Performance and safety of the device | Baseline and 12 weeks after baseline
  Users' perception of the exergaming program will be investigated by qualitative methods using short interviews or a self-made questionnaire. A total of 16 questions evaluate the rehabilitation with exergaming strategy and answers are assessed with Visual Analog Score (VAS), 0- strongly disagree, 5-strongry agree. The final score range from 0-80, where 80 indicates more positive feedback.

CONTACTS AND LOCATIONS:
Locations (1):
- COPD-Center, Gothenburg, VGR, Sweden